CLINICAL TRIAL: NCT04294862
Title: An Open-Label Study to Evaluate Tissue Distribution, Plasma Pharmacokinetics, Safety, and Tolerability After a Single Intravenous Dose of TNP-2092 in Adult Participants Undergoing Primary Total Hip or Knee Arthroplasty
Brief Title: Tissue Distribution, Pharmacokinetics, Safety, and Tolerability After a Single Dose of TNP-2092 in Participants Undergoing Primary Total Hip or Knee Arthroplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TenNor Therapeutics Limited (Industry)
Responsible Party: Sponsor
Organization: TenNor Therapeutics Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PJI001-04
Record Dates: First submitted 2020-02-25; First posted 2020-03-04 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Prosthetic Joint Infection
Keywords: TNP-2092; tissue distribution; THA; TKA; safety; PK
MeSH Terms: interventions — TNP-2092; CBR 2092

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TNP-2092 300mg IV (Experimental): TNP-2092 for injection 100mg/vial, 300mg, BID, 1 dose
  Interventions: Drug: TNP-2092

INTERVENTIONS:
Drug: TNP-2092 — TNP-2092 for injection 100mg/vial
  Other Names: CBR-2092

SUMMARY:
This study will investigate TNP-2092 distribution into joint tissues in participants undergoing a total hip arthroplasty (THA) or a total knee arthroplasty (TKA). Tissue distribution is the primary objective, and plasma pharmacokinetics (PK), safety, and tolerability are secondary objectives.

DETAILED DESCRIPTION:
This is a Phase 1, open-label study to evaluate the tissue distribution, plasma PK, safety, and tolerability after a single 300 mg intravenous (IV) dose of TNP-2092 administered before induction of anesthesia in adult participants undergoing THA or TKA. Sixteen patients who are scheduled to undergo primary THA or TKA will be enrolled.

The enrolled participants who meet the inclusion/exclusion criteria will receive the study intervention (a single 300 mg IV dose of TNP-2092) 2 hours before induction of anesthesia on Day 1. Tissue samples from bone and synovial fluid will be collected during surgery and analyzed for TNP-2092 and cefazolin concentrations. Plasma samples will be collected on Day 1 and Day 2 for PK analysis. Safety and tolerability information will be collected on Day 1 and Day 2 at the clinical center, on Day 7 by phone, and on Day 14 at a final follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all inclusion criteria are met:

1. Male or females, 18 years of age or older
2. Participants who require primary THA or TKA
3. Body mass index (BMI) >=18 kg/m2 but <=40 kg/m2
4. Capable of giving signed informed consent

Exclusion Criteria:

Participants are excluded from the study if any of the following exclusion criteria are met:

1. History or hypersensitivity or intolerability to any of the following drugs: any member of fluoroquinolones, rifamycin, cefazolin or TNP-2092
2. History of known methicillin-resistant Staphylococcus aureus (MRSA) infections
3. Presence of any surgical or medical condition that in the opinion of the principal investigator and the medical monitor that could impact the interpretation of the results of the study;
4. Evidence of significant hepatic, hematologic or immunologic disease;
5. History or evidence of severe renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Concentration of TNP-2092 in synovial fluid | 2 hours after infusion
  Concentration in ng/mL
Concentration of TNP-2092 in bone | 2 hours after infusion
  Concentration in ng/g

SECONDARY OUTCOMES:
Plasma PK of a single IV dose of TNP-2092 | pre-dose, end of infusion, 1 hours, 3 hous, 6 hours, 12 hours and 24 hours after infusion
  CTissue: Drug concentration in tissue, ng/mL
Plasma PK of a single IV dose of TNP-2092 | pre-dose, end of infusion, 1 hours, 3 hous, 6 hours, 12 hours and 24 hours after infusion
  Cmax: Peak plasma concentration,ng/mL
Plasma PK of a single IV dose of TNP-2092 | pre-dose, end of infusion, 1 hours, 3 hous, 6 hours, 12 hours and 24 hours after infusion
  Tmax: Time to maximum plasma concentration, hours
Plasma PK of a single IV dose of TNP-2092 | pre-dose, end of infusion, 1 hours, 3 hous, 6 hours, 12 hours and 24 hours after infusion
  AUC0-24: AUC versus time from time 0 to 24 hours, h*ng/mL
Rate of adverse event with TNP-2092 | Day2, Day7, Day14
  Description of adverse events as assessed by CTCAE 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopedic Institute, Philadelphia, Pennsylvania, United States